CLINICAL TRIAL: NCT00820508
Title: A Phase I Study to Evaluate the Safety and Tolerability of the Histone Deacetylase Inhibitor, CHR-2845, in Patients With Advanced or Treatment Refractory Haematological Diseases or Lymphoid Malignancies
Brief Title: Safety and Tolerability of CHR-2845 to Treat Haematological Diseases or Lymphoid Malignancies
Acronym: CHR-2845-001
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chroma Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHR-2845-001
Record Dates: First submitted 2009-01-09; First posted 2009-01-12 (Estimated); Last update posted 2011-11-28 (Estimated); Status verified 2011-11

CONDITIONS: Hematological Disease; Lymphoid Malignancies
Keywords: Haematological disease; Lymphoid malignancy; Histone deacetylase inhibitor; dose escalation
MeSH Terms: conditions — Hematologic Diseases | interventions — CHR 2845

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Oral, once daily administration of CHR-2845 to determine safety and tolerability
  Interventions: Drug: CHR-2845

INTERVENTIONS:
Drug: CHR-2845 — Once daily oral ingestion of capsules (10, 40 or 80mg), dose depending on cohort, treatment cycle of 28 days

SUMMARY:
The purpose of this study is to determine whether the histone deacetylase inhibitor CHR-2845 is tolerated in patients with haematological diseases and lymphoid malignancies.

DETAILED DESCRIPTION:
CHR-2845 is a novel type of histone deacetylase inhibitor (HDACi) for use in cancer that, in addition to having broad ranging anti-proliferative activity against transformed cells, is designed to have an increased therapeutic window against diseases which involve cells of the monocyte-macrophage lineage. There are several HDACi's in clinical development and one, SAHA (Vorinostat, Zolinza®), has recently been approved for use in the treatment of cutaneous T-cell lymphoma. CHR-2845 is a cell-permeant ester that is metabolised to give an active acid, CHR-2847, which selectively accumulates in monocytes and macrophages. This results in a 20-100 fold increase in anti-proliferative potency of CHR-2845 for monocytic over non-monocytic tumour cells. This selectivity should lead to an increased therapeutic window in haematological malignancies involving cells of the monocyte lineage (AML M4, AML M5 and CMML). In addition, there is increasing evidence that monocytes and macrophages associated with some haematological tumours (tumour-associated macrophages (TAMs)) are involved in supporting the growth and spread of the tumour. This clinical trial will focus on haematological and lymphoid malignancies with the intention of evaluating the safety and tolerability of CHR-2845. Additionally it will compare response in patients where monocytes/macrophages are important disease drivers, with the response in other patients. This will allow an early determination of the potential improvement in therapeutic window afforded by the monocyte/macrophage directed HDACi activity.

ELIGIBILITY:
Inclusion Criteria:

1. Signed, informed consent
2. Confirmed malignant haematological disease or lymphoid malignancy refractory to standard therapy or for which no standard therapy exists, including acute leukemias, MDS, CML, CLL, CMML, multiple myeloma and Non-Hodgkin's Lymphomas/Hodgkin's disease
3. Patients shall have recovered from all acute adverse effects of prior therapies, with the exception of alopecia and grade 1 neuropathy where recovery is not required
4. Adequate bone marrow, hepatic and renal function including the following:

   1. Patients with high blast counts can be included if they can be controlled by the use of hydroxyurea (500 mg -3,000 mg daily).
   2. Total bilirubin ≤ 1.5 x upper normal limit, excluding cases where elevated bilirubin can be attributed to Gilbert's Syndrome
   3. AST (SGOT), ALT (SGPT) ≤ 2.5 x upper normal limit
   4. Creatinine ≤ 1.5 x upper normal limit
5. Age ≥ 18 years
6. Performance status (PS) ≤ 2 - Eastern Cooperative Oncology Group (ECOG) scale
7. Estimated life expectancy greater than 3 months
8. Female patients with reproductive potential must have a negative serum pregnancy test within 7 days prior to start of trial. Both women and men must agree to use a medically acceptable method of contraception throughout the treatment period and for 3 months after discontinuation of treatment.

Exclusion Criteria:

1. Patients receiving anti-cancer therapy or use of other investigational agents within 21 days prior to trial entry (or a longer period depending on the defined characteristics of the agents used. Bisphosphonates for bone disease and corticosteroids are permitted provided the dose does not change during the trial. Patients must have recovered from all transient toxicity induced by prior therapy
2. Patients with co-existing active infection, graft versus host disease or serious concurrent illness
3. Patients who have failed to recover from or after a bone marrow transplantation or haematopoietic stem cell transplantation
4. The following diseases are excluded: Burkitt's lymphoma, primary effusion lymphoma, precursor B-cell lymphoblastic lymphoma, symptomatic central nervous system (CNS) lymphoma, CML blast crisis
5. Patients with significant cardiovascular disease as defined by:

   1. history of congestive heart failure requiring therapy
   2. history of angina pectoris requiring treatment or myocardial infarction within 6 months prior to trial entry
   3. presence of severe valvular heart disease
   4. presence of an atrial or ventricular arrhythmia requiring treatment
   5. Left Ventricular Ejection Fraction (LVEF) below the normal range at the study centre
   6. Uncontrolled hypertension
   7. A history of abnormal QTc intervals or an average QTc interval at screening ≥450 msec
6. Any medical or other condition that in the investigator's opinion renders the patient unsuitable for this study due to unacceptable risk
7. Psychiatric disorders or altered mental status precluding understanding of the informed consent process and/or completion of the necessary studies
8. Gastrointestinal disorders that may interfere with absorption of the study drug
9. Patients with known brain tumours or metastases
10. More than 6 prior chemotherapy regimens
11. Patients requiring growth factor support (erythropoietin, Granulocyte/monocyte Colony Stimulating Factor (GM/CSF), etc)
12. Patients requiring palliative radiotherapy within the last 4 weeks prior to study entry
13. Uncontrolled hypercalcaemia (CTCAE v3 grade 2 or higher)
14. Abnormal plasma potassium or magnesium levels (Common Terminology Criteria for Adverse Events (CTCAE) v3 grade 3 or greater) despite therapy
15. Pregnant or breast-feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2008-12; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
To determine the safety, tolerability, dose-limiting toxicities (DLT), maximum acceptable dose (MAD) and maximum tolerated dose (MTD) | 28 days

SECONDARY OUTCOMES:
To determine pharmacokinetic parameters of CHR-2845 and the active metabolite CHR-2847 | days 1 and 28

CONTACTS AND LOCATIONS:
Overall Officials: Bob Löwenberg, M.D, Principal Investigator — Erasmus Medical Center; Gert Ossenkoppele, M.D, Principal Investigator — Amsterdam UMC, location VUmc; Pierre Zachee, MD, Principal Investigator — ZNA Stuivenberg; Norbert Vey, MD, Principal Investigator — Institut Paoli-Calmettes
Locations (4):
- ZNA Stuivenberg, Antwerp, Belgium
- Institut Paoli-Calmettes, Marseille, France
- Netherlands (2):
  - VU University Medical Center, Amsterdam
  - Erasmus University Medical Center, Rotterdam

REFERENCES:
- [Derived] Ossenkoppele GJ, Lowenberg B, Zachee P, Vey N, Breems D, Van de Loosdrecht AA, Davidson AH, Wells G, Needham L, Bawden L, Toal M, Hooftman L, Debnam PM. A phase I first-in-human study with tefinostat - a monocyte/macrophage targeted histone deacetylase inhibitor - in patients with advanced haematological malignancies. Br J Haematol. 2013 Jul;162(2):191-201. doi: 10.1111/bjh.12359. Epub 2013 May 7. PMID 23647373